CLINICAL TRIAL: NCT01188135
Title: Antidepressant Adherence Via Telephonic Interactive Voice Recognition (IVR)
Brief Title: Antidepressant Adherence Via AD_IVR
Acronym: AD_IVR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MH090160 (NIH); 1R01MH090160 (NIH)
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Major Depressive Disorder
Keywords: depression; interactive voice messaging; patient persistence with antidepressant medication treatment
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interactive Voice messaging (Experimental): Participants will receive three kinds of interventions calls from the IVR phone system. (1) The first call is to orient the participant to the IVR system, ask permission to leave detailed messages in the future, and to encourage adherence in this initial period of great risk for premature discontinuation. (2) The Refill Reminder Call is to remind patients that a refill their antidepressant medications and occurs approximately 6 days before the prior dispense of medication is due to run out. (3) The "Tardy" Refill Call is made to participants for whom EMR records indicate that a scheduled refill was missed
  Interventions: Behavioral: Interactive voice messaging or Interactive voice messaging + psycho ed materials
- Usual care arm (No Intervention): usual care treatment with no interactive phone reminder calls phone
- IVR messaging w/ Psycho-ed. materials (Experimental): Participants will receive three kinds of interventions calls from the IVR phone system. (1) The first call is to orient the participant to the IVR system, ask permission to leave detailed messages in the future, and to encourage adherence in this initial period of great risk for premature discontinuation. (2) The Refill Reminder Call is to remind patients that a refill their antidepressant medications and occurs approximately 6 days before the prior dispense of medication is due to run out. (3) The "Tardy" Refill Call is made to participants for whom EMR records indicate that a scheduled refill was missed. In addition, participants will receive educational material about antidepressant medication.
  Interventions: Behavioral: Interactive voice messaging or Interactive voice messaging + psycho ed materials

INTERVENTIONS:
Behavioral: Interactive voice messaging or Interactive voice messaging + psycho ed materials — Interactive voice telephone messages reminder participants to continue to take their antidepressive medications
  Arms: IVR messaging w/ Psycho-ed. materials; Interactive Voice messaging

SUMMARY:
Antidepressants are the most frequently prescribed class of psycho¬tropic medications and the most common treatment for depression and anxiety disorders-yet patient adherence is poor and is widely viewed as contributing to reduced effectiveness. However, traditionally-delivered adherence promotion programs are complex, staff-intensive, and costly-barriers to wider adoption, implementation, and maintenance of these programs in real-world settings. Our aim is to carry out a trial of a low-cost, IT-enabled Antidepressants adherence program, specifically a direct-to-patient, automated telephone interactive voice recognition (IVR) intervention to boost patient Antidepressants persistence. We will conduct a randomized clinical trial enrolling at least 6,000 Kaiser Permanente NW Region health plan members ages 21 to 75, who had recently started on Antidepressants medications for depression and/or anxiety diagnoses. Participants will be randomized one of four arms;1. a no contact control arm, 2. a treatment as usual (TAU) control condition 3. to TAU plus the IVR automated telephone program and 4. a TAU plus the IVR automated telephone program plus receipt of psycho-education materials about antidepression medication use. Recruitment will continue for up to 18 months, with periodic participant-level follow-up assessment for the intervention participants for 40 weeks. The IVR intervention portion of the program will deliver reminder and/or tardy calls timed to projected Antidepressants refill dates. The intervention also optionally offers brief psycho-education, or transfer to a live pharmacist or the Kaiser mail refill pharmacy. The primary outcome will be the Estimated Level of Persistence with Therapy (continued us of Antidepressants medications). This will be based on prescription refill data abstracted from the Kaiser's electronic medical record (EMR). We hypothesize that participants in the IVR + psycho-education materials study arm will have a significantly higher rate of Antidepressants persistence than those in the TAU control condition ons only IRV call arms. We will also conduct cost-effectiveness analyses to assess the value-for-money (cost per depression free day gained, and cost per quality adjusted life year gained) of the IVR technology compared to TAU. Costs will include IVR development and implementation as well as EMR-derived healthcare utilization data (visits, medications, etc.), augmented with participant report of out-of-plan services.

DETAILED DESCRIPTION:
Antidepressants (AD) are the most frequently prescribed class of psycho-tropic medications and the most common treatment for depression and anxiety disorders-yet patient adherence is poor and is widely viewed as contributing to reduced effectiveness. Fortunately, AD adherence can be improved via interventions consistent with the Chronic Care Model (CCM). However, traditionally-delivered adherence promotion programs are complex, staff-intensive, and costly-barriers to wider adoption, implementation, and maintenance of these programs in real-world settings. Our aim is to carry out a trial of a low-cost, IT-enabled AD adherence program, specifically a direct-to-patient, automated telephone interactive voice recognition (IVR) intervention to boost patient AD persistence. This intervention is consistent with the Chronic Care Model but is much more amenable to widespread dissemination over a large population. In an initial startup period the investigators will adapt and pilot existing IVR adherence calls and scripts, informed by formative focus groups and interviews with key informants (patients, providers). Following this, the investigators will conduct a pragmatic, randomized clinical trial at approximately 6,000 HMO members ages 21 to 75, recently started on an incident course of AD medications for associated unipolar depression and/or anxiety diagnoses. Participants will be randomized (1:1:1:1); 1. a no contact control arm, 2. a treatment as usual (TAU) control condition 3. to TAU plus the IVR automated telephone program and 4. a TAU plus the IVR automated telephone program plus receipt of psycho-education materials about antidepression medication use. Recruitment will continue for up to 18 months, with periodic participant-level follow-up for 40 weeks. The two IVR interventions will deliver reminder and/or tardy calls timed to projected AD refill dates. The intervention arms also optionally offers transfer to a live pharmacist or the HMO mail refill pharmacy. The primary outcome will be the Estimated Level of Persistence with Therapy (ELPT) for ADs, based on prescription refill data abstracted from the HMO's electronic medical record (EMR). We hypothesize that participants in the IVR study plus psycho-ed. arm will have a significantly higher rate of AD persistence than those in the TAU control condition or IVR only. Secondary medication adherence outcomes include continuous measure of medication acquisition (CMA) and continuous measure of medication gaps (CMG). Other secondary outcomes include self-report depression and anxiety symptoms, general health status, patient and provider satisfaction, and healthcare costs and usage. We will also conduct cost-effectiveness analyses (CEA) to assess the value-for-money (cost per depression free day gained, and cost per quality adjusted life year gained) of the IVR technology compared to TAU. Costs will include IVR development and implementation as well as EMR-derived healthcare utilization data (visits, medications, etc.), augmented with participant report of out-of-plan services. Finally, evaluative qualitative interviews will be conducted with key stakeholders to identify barriers/facilitators of intervention implementation-keys for future dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be Kaiser Permanente NW Region health plan members ages of 21 and 75 and be members for at least 6 months prior to the initial antidepressive medications dispense.
* Participants must have an EMR chart diagnosis or presenting complaint of a unipolar mood diagnosis, anxiety disorder, or any subclinical or "not otherwise categorized" (NOC) variant of these.
* The participants' providers must give permission to study staff for their patients' enrollment in the study. There must be no indication of pending HMO disenrollment in the membership data.
* Participants must have an initial dispense of an antidepressant medication, with no dispense of any of these agents in the prior 6 months.

Exclusion Criteria:

* Participants must have no EMR chart diagnosis that is likely to impair participant ability to complete evaluations or take part in the intervention. These include psychiatric diagnoses such as bipolar disorder I (BP II is acceptable), schizophrenia, schizo-affective disorder, or similar diagnoses indicating psychosis.
* The investigators will also exclude individuals with any chart diagnosis indicating significant intellectual impairment, such as any dementia disorder, mental retardation, or profound developmental disorder such as autism.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6058 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Participants in the IVR study arm will have a significantly higher rate of AD persistence (ELPT) than those in the TAU control condition | assessments at 4, 8,12 and 40 weeks
  A randomized controlled trial of adult members of a (HMO) starting an incident episode of antidepressant treatment, (a) nocontact control,(b) treatment as usual (TAU) versus (c) TAU plus the IVR automated telephone adherence program, (d)TAU plus the IVR automated telephone adherence program plus mailed psycho-education materials. The primary outcome will be antidepressant persistence, operationalized as the Estimated Level of Persistence with Therapy. Secondary outcomes will include patient and provider satisfaction, healthcare utilization, and patient self-reported depression and anxiety.

SECONDARY OUTCOMES:
cost-effectiveness analyses | at the end of week 40
  We will also conduct cost-effectiveness analyses comparing the arms of the study. We will employ healthcare utilization data (visits, medications, etc.) obtained from the electronic medical record, augmented with participant report of out-of-plan healthcare services. These will compare study conditions on the cost to achieve units of improvement in depression free days and quality-adjusted life years. We expect that costs per unit of improvementfor the IVR intervention will be within standard boundaries of decision-makers willingness to pay.

CONTACTS AND LOCATIONS:
Overall Officials: Greg N Clarke, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States